CLINICAL TRIAL: NCT01754571
Title: Cognitive Behavior Therapy in Patients With Medication Overuse
Brief Title: CBT in Patients With Medication Overuse Headache
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 101041-E
Record Dates: First submitted 2012-08-15; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Medication Overuse Headache
Keywords: medication overuse headache
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CBT treatment (Experimental)
  Interventions: Behavioral: Cognitive behavior therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Behavior therapy, including Relaxation, cognitive rebuilding.

SUMMARY:
According to the definition from International Headache Society, medication overuse headache (MOH) is diagnosed when patients takes painkillers for more than 10 or 15 days per month (depending on what kind of painkillers being used), for more than 3 months, which results in the deterioration of headache. The treatments of MOH include preventive medication of headache and withdrawal of the overused painkillers. Other than the simple oral advice, some researchers recommended non-pharmacological methods. Pryse-Phillips et al. (1998) reviewed the the treatment of migraine and suggested that biofeedback, relaxation, cognitive behavior therapy (CBT), psychological therapy, hypnosis and physical treatment are effective. Researches also point out CBT is effective on withdrawing medication in patients with MOH (Kroner-Herwig, 2009). Lake (2006) reported that behavioural therapy maybe an adjunct therapy to preventive medication to reduce the relapse rate of medication overuse.

The purpose of this study is to confirm the effect of CBT in patients with MOH. The target is to reduce the frequency of headache and use of painkillers. Patients could benefit from the education and relaxation training during CBT to cope with headache and reduce the use of painkillers.

The research will recruit 60 patients with MOH at Neurology Clinics, Far Eastern Memorial Hospital. They will be separated into two groups, 30 in control group and the other 30 in the experimental group. Education of MOH, relaxation and cognitive restructuring would be included in the four weeks training program. The training program is under the supervision of a neurologist from Far Eastern Memorial Hospital and a psychology professor from Fu Jen Catholic University. The control group will accept four weeks telephone interview to confirm their headache diary including the frequency of headache and use of painkillers. The frequency of headache and medication use will be used for analyzing the effect of CBT.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Medication overuse headache

Exclusion Criteria:

* other type headache

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan